CLINICAL TRIAL: NCT01911338
Title: EFFECT OF REAL-TIME FEEDBACK THROUGH INERTIAL SENSORS IN LEARNING POSTEROANTERIOR THORACIC MANIPULATION
Brief Title: Inertial Sensors Used to Learn Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, PhD, University of Malaga
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: ACuesta07072013
Record Dates: First submitted 2013-07-23; First posted 2013-07-30 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2013-07

CONDITIONS: Medical Education
Keywords: Spinal Manipulation; Teaching; Thoracic Vertebrae; Feedback

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real Time Feedback (Experimental): Before beginning practice, one of the teachers performed the manipulation and explained the graph parameters as real-time feedback to consider when interpreting the graph, leaving the graphic as the benchmark execution
  Interventions: Device: Real Time Feedback
- Tradicional Learning Method (Active Comparator): Two expert teachers in manual therapy provided indications and corrections to the group with a teacher - student ratio of 1:8
  Interventions: Device: Traditional Learning Method

INTERVENTIONS:
Device: Real Time Feedback — Before beginning practice, one of the teachers performed the manipulation and explained the graph parameters as real-time feedback to consider when interpreting the graph, leaving the graphic as the benchmark execution
  Arms: Real Time Feedback
Device: Traditional Learning Method — Two expert teachers in manual therapy provided indications and corrections to the group with a teacher - student ratio of 1:8.
  Arms: Tradicional Learning Method

SUMMARY:
* Background Context: no studies have been identified to analyse the effect of real time feedback (using inertial sensors) on physiotherapy students learning the art of posterior-anterior thoracic manipulation (PATM).
* Purpose: to study the effect caused by real-time feedback on the learning process for PATM, comparing two undergraduate physiotherapy student groups. Hypothesis: significant differences will exist in the execution parameters of manipulation among students receiving real-time feedback versus those who do not.
* Study Design/Setting: longitudinal, pre-post intervention.
* Patient Sample: Sixty-one undergraduate physiotherapy students were divided randomly into two groups, G1 (n = 31) (group without feedback in real time) and G2 (n = 30) (group with real-time feedback).
* Outcome Measures: time, displacement and velocity and improvement (only between groups) to reach maximum peak, to reach minimum peak from maximum peak, total manipulation time.
* Methods: two groups of physiotherapy students learned PATM, one using a traditional method and the other using real-time feedback (inertial sensor). Measures were obtained pre- and post-intervention. Intragroup pre- and post-intervention and intergroup post-intervention scores were calculated. An analysis of the measures' stability was developed through an ICC (1,2).
* Results: the values of ICC ranged from 0.881 to 0.997. Statistically significant differences were found in all variables analysed (intra- and inter-group) in favour of G2.
* Conclusions: the learning process for posterior-anterior thoracic manipulation is facilitated when the student receives real-time feedback.

ELIGIBILITY:
Inclusion Criteria:

* Participants did not have any training in manual therapy techniques, especially those involving a high velocity, low amplitude execution.

Exclusion Criteria:

* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change from displacement maximum peak (seconds) | baseline; post-education; 24 weeks follow up
  An instrumented manikin (Resusci Anne Full Body with signal box, Laerdal Medical AS) joined an inertial sensor (Inertial Cube (Intersense Inc, USA)) was used to register the physical parameters during execution of the PATM. The inertial sensor was placed in the middle of the thoracic spine, placing hands immediately below the sensor. The manikin has a ribcage with a deformation capacity similar to that of a human thorax. This option was chosen to minimize the power variation when comparing differences in parameters between different groups of students. The inclusion criteria used were that they did not have any training in manual therapy techniques, especially those involving a high velocity, low amplitude execution.
Change from Time to reach maximum peak (seconds) | baseline; post-education; 24 weeks follow up
  An instrumented manikin (Resusci Anne Full Body with signal box, Laerdal Medical AS) joined an inertial sensor (Inertial Cube (Intersense Inc, USA)) was used to register the physical parameters during execution of the PATM. The inertial sensor was placed in the middle of the thoracic spine, placing hands immediately below the sensor. The manikin has a ribcage with a deformation capacity similar to that of a human thorax. This option was chosen to minimize the power variation when comparing differences in parameters between different groups of students. The inclusion criteria used were that they did not have any training in manual therapy techniques, especially those involving a high velocity, low amplitude execution.
Change from Displacement between maximum and minimum peak (milimitres) | baseline; post-education; 24 weeks follow up
  An instrumented manikin (Resusci Anne Full Body with signal box, Laerdal Medical AS) joined an inertial sensor (Inertial Cube (Intersense Inc, USA)) was used to register the physical parameters during execution of the PATM. The inertial sensor was placed in the middle of the thoracic spine, placing hands immediately below the sensor. The manikin has a ribcage with a deformation capacity similar to that of a human thorax. This option was chosen to minimize the power variation when comparing differences in parameters between different groups of students. The inclusion criteria used were that they did not have any training in manual therapy techniques, especially those involving a high velocity, low amplitude execution.
Change from Total manipulation time (seconds) | baseline; post-education; 24 weeks follow up
  An instrumented manikin (Resusci Anne Full Body with signal box, Laerdal Medical AS) joined an inertial sensor (Inertial Cube (Intersense Inc, USA)) was used to register the physical parameters during execution of the PATM. The inertial sensor was placed in the middle of the thoracic spine, placing hands immediately below the sensor. The manikin has a ribcage with a deformation capacity similar to that of a human thorax. This option was chosen to minimize the power variation when comparing differences in parameters between different groups of students. The inclusion criteria used were that they did not have any training in manual therapy techniques, especially those involving a high velocity, low amplitude execution.
Change from Velocity to reach maximum peak (degrees per second) | baseline; post-education; 24 weeks follow up
  An instrumented manikin (Resusci Anne Full Body with signal box, Laerdal Medical AS) joined an inertial sensor (Inertial Cube (Intersense Inc, USA)) was used to register the physical parameters during execution of the PATM. The inertial sensor was placed in the middle of the thoracic spine, placing hands immediately below the sensor. The manikin has a ribcage with a deformation capacity similar to that of a human thorax. This option was chosen to minimize the power variation when comparing differences in parameters between different groups of students. The inclusion criteria used were that they did not have any training in manual therapy techniques, especially those involving a high velocity, low amplitude execution.
Change from Time to reach peak minimum from maximum peak (seconds) | baseline; post-education; 24 weeks follow up
  An instrumented manikin (Resusci Anne Full Body with signal box, Laerdal Medical AS) joined an inertial sensor (Inertial Cube (Intersense Inc, USA)) was used to register the physical parameters during execution of the PATM. The inertial sensor was placed in the middle of the thoracic spine, placing hands immediately below the sensor. The manikin has a ribcage with a deformation capacity similar to that of a human thorax. This option was chosen to minimize the power variation when comparing differences in parameters between different groups of students. The inclusion criteria used were that they did not have any training in manual therapy techniques, especially those involving a high velocity, low amplitude execution.
Change from Velocity to reach minimum peak from maximum peak (degress/second) | baseline; post-education; 24 weeks follow up
  An instrumented manikin (Resusci Anne Full Body with signal box, Laerdal Medical AS) joined an inertial sensor (Inertial Cube (Intersense Inc, USA)) was used to register the physical parameters during execution of the PATM. The inertial sensor was placed in the middle of the thoracic spine, placing hands immediately below the sensor. The manikin has a ribcage with a deformation capacity similar to that of a human thorax. This option was chosen to minimize the power variation when comparing differences in parameters between different groups of students. The inclusion criteria used were that they did not have any training in manual therapy techniques, especially those involving a high velocity, low amplitude execution.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel González-Sánchez, PT, PhD, Principal Investigator — University of Malaga; Yves Lenfant, PT, Principal Investigator — University of Malaga